CLINICAL TRIAL: NCT06244394
Title: A Retrospective Study to Establish a Prediction Model for Radiation-induced Brain Damage in Nasopharyngeal Carcinoma Patients Based on Pretreatment Imaging and Radiotherapy Data
Brief Title: Retrospective Study on the Prediction of Radiation-induced Brain Injury in Patients With Nasopharyngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Lirong Wu, Associate chiefphysician, Jiangsu Cancer Institute & Hospital
Other Study IDs: RTLI prediction model
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Nasopharyngeal Carcinoma; Radiation-Induced Temporal Lobe Injury
Keywords: radiomics; machine learning; deep learning
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NPC patients with RTLI after IMRT: nasopharyngeal carcinoma patients with radiation-induced temporal lobe injury after intensity-modulated radiation therapy
  Interventions: Radiation: intensity-modulated radiotherapy
- NPC patients without RTLI after IMRT: nasopharyngeal carcinoma patients without radiation-induced temporal lobe injury after intensity-modulated radiation therapy
  Interventions: Radiation: intensity-modulated radiotherapy

INTERVENTIONS:
Radiation: intensity-modulated radiotherapy — All patients were staged according to the 8th edition of the TNM classification by the American Joint Committee on Cancer/Union for International Cancer Control and received a standardized treatment regimen including IMRT and concurrent or adjuvant chemotherapy. Inverse IMRT treatment planning was performed on a Varian Inspiration Platform (version 10.0), using the simultaneous integrated boost technique. The prescribed doses were 68-75 Gy to the PTV of the GTVnx in 32-34 fractions; 64-75 Gy to the PTV of the GTVnd in 32-34 fractions; 60 Gy to the PTV of CTV1 in 32 fractions; and 50 Gy to the PTV of CTV2 in 28 fractions. All patients were given one fraction daily 5 days a week. The dose-volume-histograms (DVHs) of the organs at risk were evaluated as described in the radiation therapy oncology group (RTOG) 0225 protocol to prevent violation of the tolerance limits.

SUMMARY:
Radiation therapy has become the preferred treatment for nasopharyngeal cancer due to the sensitivity of nasopharyngeal carcinoma to radiation. However, even with the use of intensity-modulated radiation therapy (IMRT), radiation-induced temporal lobe injury (RTLI) can be a severe complication. Patients with RTLI may experience long-term memory loss, personality changes, physical dysfunctions, and other symptoms, which seriously impair their quality of life and long-term prognosis. Currently, the diagnosis of RTLI primarily relies on clinical symptoms and imaging examinations such as computed tomography (CT) and conventional MRI. However, these methods only enable the diagnosis of RTLI at a late stage when it is irreversible and cannot be effectively treated. Therefore, the early identification or individualized prediction of RTLI after IMRT holds exceptional importance for improving the quality of life in nasopharyngeal carcinoma patients.

The exact mechanism of RTLI remains unclear. Many clinical covariates have been proven to be associated with RTLI in NPC patients, including stage, age, and dosimetric parameters. In addition, it was reported that each patient's temporal lobe exhibits unique genetic susceptibility to radiation exposure. In this study, we aim to predict the occurrence of RTLI by analyzing clinical factors and heterogeneity of temporal lobe tissue prior to irradiation. Finally, we want to construct and validate a prediction model for RLTI, which can support clinician decision-making in developing individualized treatment plans and providing preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* (1) pathological confirmation of NPC; (2) receipt of IMRT; (3) nasopharynx-neck MRI within 2 weeks before antineoplastic treatment

Exclusion Criteria:

* (1) temporal lobe invasion; (2) with central nervous system diseases except RTLI; (3) receiving additional radiation after IMRT; (4) incomplete clinical or imaging data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: nasopharyngeal carcinoma paients who recieved intensity-modulated radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
NPC patients with RTLI | three years
  Patients with nasopharyngeal cancer who were diagnosed with radiation-induced brain injury during follow-up period
NPC patients without RTLI | three years
  Patients with nasopharyngeal cancer who were not diagnosed with radiation-induced

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No